CLINICAL TRIAL: NCT00321763
Title: Demonstrate the Lot-to-lot Consistency of 3 Consecutive Production Lots of an Adjuvanted Influenza Vaccine Candidate and Evaluate the Safety of an Adjuvanted Influenza Vaccine Candidate Versus Fluarix™ Administered Intramuscularly in Elderly
Brief Title: Study to Demonstrate the Lot-to-lot Consistency and to Evaluate the Safety of an Adjuvanted Influenza Vaccine Candidate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107192; 107214 (Other: GSK)
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: Influenza; Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (5):
- GSK1247446A Lot 1 Group (Experimental): Subjects aged 60 years or older at the time of vaccination received 1 dose of Lot 1 GSK1247446A vaccine adjuvanted with AS03 at Day 0. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Candidate Influenza Vaccine GSK1247446A - 3 different formulations
- GSK1247446A Lot 2 Group (Experimental): Subjects aged 60 years or older at the time of vaccination received 1 dose of Lot 2 GSK1247446A vaccine adjuvanted with AS03 at Day 0. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Candidate Influenza Vaccine GSK1247446A - 3 different formulations
- GSK1247446A Lot 3 Group (Experimental): Subjects aged 60 years or older at the time of vaccination received 1 dose of Lot 3 GSK1247446A vaccine adjuvanted with AS03 at Day 0. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Candidate Influenza Vaccine GSK1247446A - 3 different formulations
- GSK1247446A Pooled Group (Experimental): Subjects aged 60 years or older at the time of vaccination received 1 dose of Lot 1, 2 or 3 GSK1247446A vaccines adjuvanted with AS03 at Day 0. The vaccines were administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Candidate Influenza Vaccine GSK1247446A - 3 different formulations
- Fluarix Group (Active Comparator): Subjects aged 60 years or older at the time of vaccination received 1 dose of FluarixTM vaccine adjuvanted with AS03 at Day 0. The vaccines were administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix TM

INTERVENTIONS:
Biological: Candidate Influenza Vaccine GSK1247446A - 3 different formulations — Single dose, Intramuscular injection
  Arms: GSK1247446A Lot 1 Group; GSK1247446A Lot 2 Group; GSK1247446A Lot 3 Group; GSK1247446A Pooled Group
Biological: Fluarix TM — Single dose, Intramuscular injection
  Arms: Fluarix Group

SUMMARY:
The purpose of this phase IIb study is to demonstrate the consistency of three lots of an adjuvanted influenza vaccine candidate and to evaluate the safety of this vaccine compared to Fluarix™ administered intramuscularly in elderly aged 60 years old and above.

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A male or female age 60 years or older at the time of the vaccination.
* Subjects who the investigator believes can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the administration of the study vaccine, or planned use during the study period.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within three months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to 30 days after vaccination.
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of confirmed influenza infection within the last 12 months.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s)
* Acute disease at the time of enrolment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3124 (Actual)
Dates: Start 2006-04-27; Primary Completion 2006-07-01 (Actual); Study Completion 2006-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- GSK Investigational Site, Tartu, Estonia
- France (9):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Gières
  - GSK Investigational Site, Lagord
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Toulouse
- Germany (14):
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Marktl, Bavaria
  - GSK Investigational Site, Oberaudorf, Bavaria
  - GSK Investigational Site, Ketzin, Brandenburg
  - GSK Investigational Site, Koenigslutter, Lower Saxony
  - GSK Investigational Site, Tostedt, Lower Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Kamenz, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Weißenberg, Saxony
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
- Greece (8):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Goudi / Athens
  - GSK Investigational Site, Haidari
  - GSK Investigational Site, Marousi
  - GSK Investigational Site, Nikaia Piraeus
  - GSK Investigational Site, Orestiáda
  - GSK Investigational Site, Papagos/Athens
  - GSK Investigational Site, Thessaloniki
- Norway (4):
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Paradis
  - GSK Investigational Site, Stavanger
- Russia (3):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Yekaterinburg
- United Kingdom (7):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Edgbaston, Birmingham
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Waterloo, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 107192 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107192 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107192 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107192 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107192 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | Fluarix Group
Started | 850 | 850 | 854 | 570
Completed | 844 | 848 | 848 | 565
Not Completed | 6 | 2 | 6 | 5
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | Fluarix Group | Total
Number analyzed (Participants) | 850 | 850 | 854 | 570 | 3124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (6.17) | 68.8 (6.43) | 68.7 (6.54) | 68.3 (6.15) | 68.6 (6.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 475 | 451 | 479 | 340 | 1745
  Male | 375 | 399 | 375 | 230 | 1379

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 3 influenza strains assessed were A/New Caledonia, A/New York and B/Malaysia. The seropositivity cut-off assay was 1:10. The results for the GSK1247446A Lot 1, 2, 3 and Pooled Groups are the primary efficacy variables.
Time Frame: At Days 0 and 21
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning Immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 494 | 494 | 499 | 1487 | 106
titers
  A/New Caledonia, Day 0 [N=494;494;499;1487;106] | 26.7 [24.0 to 29.7] | 28.5 [25.6 to 31.7] | 28.6 [25.7 to 31.8] | 27.9 [26.2 to 29.7] | 25.7 [20.4 to 32.3]
  A/New Caledonia, Day 21 [N=492;488;492;1472;106] | 121.4 [108.9 to 135.3] | 119.1 [107.5 to 132.0] | 133.8 [120.4 to 148.8] | 124.6 [117.3 to 132.4] | 130.6 [100.3 to 170.1]
  A/New York, Day 0 [N=494;494;499;1487;106] | 24.2 [21.6 to 27.0] | 23.9 [21.4 to 26.7] | 24.3 [21.6 to 27.3] | 24.1 [22.6 to 25.7] | 26.2 [20.5 to 33.5]
  A/New York, Day 21 [N=492;488;492;1472;106] | 189.3 [168.3 to 213.0] | 192.3 [171.7 to 215.5] | 187.3 [167.5 to 209.5] | 189.6 [177.5 to 202.6] | 110.9 [85.0 to 144.7]
  B/Malaysia, Day 0 [N=494;494;499;1487;106] | 29.6 [26.4 to 33.1] | 29.7 [26.7 to 33.1] | 31.8 [28.3 to 35.6] | 30.3 [28.4 to 32.4] | 27.7 [21.5 to 35.8]
  B/Malaysia, Day 21 [N=492;488;492;1472;106] | 243.0 [218.4 to 270.2] | 229.9 [208.3 to 253.7] | 238.7 [216.5 to 263.3] | 237.1 [223.7 to 251.4] | 167.0 [131.6 to 211.8]

2. Primary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 3 assessed influenza strains were A/New Caledonia, A/New York and B/Malaysia. The results for the GSK1247446A Lot 1, 2, 3 and Pooled Groups are the primary efficacy variables.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 491 | 487 | 492 | 1470 | 106
subjects
  A/New Caledonia, Day 21 | 214 | 205 | 233 | 652 | 47
  A/New York, Day 21 | 308 | 309 | 313 | 930 | 49
  B/Malaysia, Day 21 | 333 | 317 | 326 | 976 | 59

3. Primary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 3 assessed influenza strains were A/New Caledonia, A/New York and B/Malaysia. The results for the GSK1247446A Lot 1, 2, 3 and Pooled Groups are the primary efficacy variables.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 494 | 494 | 499 | 1487 | 106
subjects
  A/New Caledonia, Day 0 [N=494;494;499;1487;106] | 221 | 220 | 229 | 670 | 46
  A/New Caledonia, Day 21 [N=491;487;492;1470;106] | 439 | 433 | 454 | 1326 | 94
  A/New York, Day 0 [N=494;494;499;1487;106] | 197 | 201 | 200 | 598 | 47
  A/New York, Day 21 [N=491;487;492;1470;106] | 451 | 447 | 454 | 1352 | 89
  B/Malaysia, Day 0 [N=494;494;499;1487;106] | 240 | 230 | 236 | 706 | 52
  B/Malaysia, Day 21 [N=491;487;492;1470;106] | 474 | 475 | 481 | 1430 | 97

4. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 3 assessed influenza strains were A/New Caledonia, A/New York and B/Malaysia. The results for the GSK1247446A Lot 1, 2, 3 and Pooled Groups are the primary efficacy variables.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 491 | 487 | 492 | 1470 | 106
fold increase
  A/New Caledonia, Day 21 | 4.6 [4.0 to 5.2] | 4.2 [3.7 to 4.7] | 4.7 [4.1 to 5.4] | 4.5 [4.2 to 4.8] | 5.1 [3.7 to 7.1]
  A/New York, Day 21 | 7.9 [6.9 to 9.0] | 7.9 [7.0 to 9.1] | 7.7 [6.8 to 8.8] | 7.8 [7.3 to 8.5] | 4.2 [3.2 to 5.5]
  B/Malaysia, Day 21 | 8.2 [7.2 to 9.3] | 7.6 [6.8 to 8.5] | 7.6 [6.7 to 8.6] | 7.8 [7.3 to 8.4] | 6.0 [4.6 to 7.9]

5. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms.
Description: Assessed solicited local symptoms were ecchymosis, pain, redness and swelling at injection site. Any = incidence of a particular symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling/ecchymosis = redness/swelling/ecchymosis spreading beyond 50 millimeters (mm) of the injection site. All solicited local symptoms were assessed by the investigator as being related to study vaccination.
Time Frame: During the 7-day (Days 0-6) post vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with a documented dose and with symptom sheets completed .
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 847 | 850 | 851 | 2548 | 568
subjects
  Any Ecchymosis | 22 | 34 | 30 | 86 | 17
  Ecchymosis > 50 mm | 1 | 2 | 3 | 6 | 0
  Any Pain | 470 | 449 | 456 | 1375 | 170
  Grade 3 Pain | 9 | 13 | 13 | 35 | 3
  Any Redness | 324 | 297 | 338 | 959 | 162
  Redness > 50 mm | 103 | 80 | 115 | 298 | 17
  Any Swelling | 241 | 208 | 238 | 687 | 87
  Swelling > 50 mm | 54 | 46 | 59 | 159 | 5

6. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache, muscle aches and shivering. Any = incidence of a particular symptom regardless of grade intensity or relationship with the study vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0°C. Related = symptom considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During the 7-day (Days 0-6) post vaccination period
Population: as for outcome 5
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 847 | 850 | 852 | 2549 | 568
subjects
  Any Arthralgia | 130 | 133 | 133 | 396 | 47
  Grade 3 Arthralgia | 9 | 10 | 12 | 31 | 2
  Related Arthralgia | 69 | 90 | 85 | 244 | 29
  Any Fatigue | 251 | 210 | 233 | 694 | 101
  Grade 3 Fatigue | 13 | 17 | 11 | 41 | 4
  Related Fatigue | 156 | 143 | 144 | 443 | 53
  Fever ≥ 37.5°C | 45 | 54 | 44 | 143 | 2
  Fever > 39.0°C | 0 | 3 | 1 | 4 | 0
  Related Fever | 35 | 34 | 28 | 97 | 1
  Any Headache | 182 | 167 | 182 | 531 | 77
  Grade 3 Headache | 8 | 11 | 8 | 27 | 3
  Related Headache | 100 | 109 | 111 | 320 | 38
  Any Muscle aches | 254 | 234 | 245 | 733 | 79
  Grade 3 Muscle aches | 8 | 13 | 17 | 38 | 0
  Related Muscle aches | 159 | 160 | 156 | 475 | 46
  Any Shivering | 92 | 93 | 90 | 275 | 28
  Grade 3 Shivering | 8 | 11 | 9 | 28 | 0
  Related Shivering | 51 | 62 | 45 | 158 | 13

7. Primary Outcome: Number of Subjects With New Onset of Chronic Diseases (NOCDs).
Description: NOCDs include conditions such as diabetes, autoimmune disease, asthma, allergies etc. This table includes rare events, defined as events with an occurrence rate of 0.1 % and belonging to the NOCDs.
Time Frame: From Day 0 to Day 180
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 850 | 850 | 854 | 2554 | 570
subjects | 3 | 3 | 2 | 8 | 1

8. Primary Outcome: Number of Subjects With Medically Significant Conditions (MSCs).
Description: MSCs were defined as conditions prompting emergency room visits or physician visits that were not related to common diseases or routine visits. This table includes rare events, defined as events with an occurrence rate of 0.1 % and belonging to the MSCs.
Time Frame: From Day 0 to Day 180
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 850 | 850 | 854 | 2554 | 570
subjects | 70 | 69 | 72 | 211 | 52

9. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = unsolicited AE that prevented normal activity Related = unsolicited AE assessed by the investigator as related to the vaccination. This table includes rare events, defined as events with an occurrence rate of 0.1 % and belonging to the AEs.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 850 | 850 | 854 | 2554 | 570
subjects
  Subjects with any AE(s) | 133 | 150 | 162 | 445 | 109
  Subjects with any Grade 3 AE(s) | 11 | 14 | 15 | 40 | 10
  Subjects with any related AE(s) | 47 | 57 | 65 | 169 | 16

10. Primary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any = any SAE regardless of intensity or relationship to vaccination. Related (REL) = SAE assessed by the investigator as related to the vaccination.
Time Frame: During the entire study period (Days 0-180)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Number analyzed (Participants) | 850 | 850 | 854 | 2554 | 570
subjects
  Any SAE(s), Days 0-29 [N=850;850;854;2554;570] | 4 | 4 | 3 | 11 | 4
  REL SAE(s), Days 0-29 [N=850;850;854;2554;570] | 0 | 0 | 0 | 0 | 0
  Any SAE(s), Days 30-180 [N=844;848;848;2540;565] | 26 | 20 | 20 | 66 | 17
  REL SAE(s), Days 30-180 [N=844;848;848;2540;565] | 0 | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAE(s): during the entire study period (Day 0 - Day 180); Solicited local and general symptoms: during the 7-day (Days 0-6) follow-up period after vaccination, Unsolicited AE(s): during the 30-day follow-up period (Days 0 to 29) after vaccination.
Arm/Group | GSK1247446A Lot 1 Group | GSK1247446A Lot 2 Group | GSK1247446A Lot 3 Group | GSK1247446A Pooled Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 30/850 | 24/850 | 23/854 | 77/2554 | 21/570
Other Adverse Events (participants affected / at risk) | 653/850 | 636/850 | 634/854 | 1923/2554 | 321/570
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK1247446A Lot 1 Group (N=850) | GSK1247446A Lot 2 Group (N=850) | GSK1247446A Lot 3 Group (N=854) | GSK1247446A Pooled Group (N=2554) | Fluarix Group (N=570)
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Abdominal pain (General disorders) | 0 | 1 | 0 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Retinal artery embolism (Eye disorders) | 0 | 1 | 0 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Retinal detachment (Eye disorders) | 0 | 1 | 0 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 — During the 30-day (Days 0 to 29) post vaccination period.
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 — During the 30-day (Days 0 to 29) post vaccination period.
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 — During the 30-day (Days 0 to 29) post vaccination period.
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 — During the 30-day (Days 0 to 29) post vaccination period.
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 — During the 30-day (Days 0 to 29) post vaccination period.
Syncope (Nervous system disorders) | 2/844 | 2/848 | 1/848 | 5/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Angina pectoris (Cardiac disorders) | 4/844 | 0/848 | 0/848 | 4/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Chest pain (General disorders) | 0/844 | 1/848 | 1/848 | 2/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Cerebrovascular accident (Nervous system disorders) | 1/844 | 1/848 | 0/848 | 2/2540 | 2/565 — During the post vaccination period between Days 30 and 180.
Cholelithiasis (Hepatobiliary disorders) | 2/844 | 0/848 | 0/848 | 2/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Circulatory collapse (Vascular disorders) | 1/844 | 0/848 | 1/848 | 2/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Constipation (Gastrointestinal disorders) | 0/844 | 0/848 | 2/848 | 2/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Coronary artery disease (Cardiac disorders) | 0/844 | 2/848 | 0/848 | 2/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Femoral neck fracture (Injury, poisoning and procedural complications) | 0/844 | 0/848 | 2/848 | 2/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/844 | 1/848 | 1/848 | 2/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Bile duct stone (Hepatobiliary disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Colonic polyp (Gastrointestinal disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Hip fracture (Injury, poisoning and procedural complications) | 0/844 | 0/848 | 1/848 | 1/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Acute myocardial infarction (Cardiac disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Anaemia (Blood and lymphatic system disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Ankle fracture (Injury, poisoning and procedural complications) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Aortic stenosis (Vascular disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Cardiovascular disorder (Cardiac disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Cerebral infarction (Nervous system disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Cholecystitis infective (Infections and infestations) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Completed suicide (Psychiatric disorders) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Diverticulitis (Infections and infestations) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Excoriation (Injury, poisoning and procedural complications) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Foot deformity (Musculoskeletal and connective tissue disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Forearm fracture (Injury, poisoning and procedural complications) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Foreign body trauma (Injury, poisoning and procedural complications) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Gastritis (Gastrointestinal disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
General physical health deterioration (General disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Hyperlipidaemia (Metabolism and nutrition disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Hyperthyroidism (Endocrine disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Iliac artery stenosis (Vascular disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Nephrolithiasis (Renal and urinary disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Nephrotic syndrome (Renal and urinary disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Pancreatitis (Gastrointestinal disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Peripheral vascular disorder (Vascular disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Pneumonia (Infections and infestations) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Scoliosis (Musculoskeletal and connective tissue disorders) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Stress (Psychiatric disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Suicide attempt (Psychiatric disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Tachyarrhythmia (Cardiac disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Tachycardia paroxysmal (Cardiac disorders) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Trigeminal neuralgia (Nervous system disorders) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Acute coronary syndrome (Cardiac disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Aortic aneurysm (Vascular disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Arrhythmia (Cardiac disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Arteriosclerosis coronary artery (Cardiac disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Gallstone ileus (Gastrointestinal disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Hypertension (Vascular disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Pyrexia (General disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Small intestinal perforation (Gastrointestinal disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565
Uterine polyp (Reproductive system and breast disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Cardiac failure (Cardiac disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Oedema (General disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Hepatorenal failure (Hepatobiliary disorders) | 1/844 | 0/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Myocardial infarction (Cardiac disorders) | 0/844 | 1/848 | 0/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Diabetic gangrene (Infections and infestations) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Road traffic accident (Injury, poisoning and procedural complications) | 0/844 | 0/848 | 1/848 | 1/2540 | 0/565 — During the post vaccination period between Days 30 and 180.
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
Thrombotic stroke (Nervous system disorders) | 0/844 | 0/848 | 0/848 | 0/2540 | 1/565 — During the post vaccination period between Days 30 and 180.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A Lot 1 Group (N=850) | GSK1247446A Lot 2 Group (N=850) | GSK1247446A Lot 3 Group (N=854) | GSK1247446A Pooled Group (N=2554) | Fluarix Group (N=570)
Pain (General disorders) | 470 | 449 | 456 | 1375 | 170
Redness (General disorders) | 324 | 297 | 338 | 959 | 162
Swelling (General disorders) | 241 | 208 | 238 | 687 | 87
Arthralgia (General disorders) | 130 | 133 | 133 | 396 | 47
Fatigue (General disorders) | 251 | 210 | 233 | 694 | 101
Fever (General disorders) | 45 | 54 | 44 | 143 | 2
Headache (General disorders) | 182 | 167 | 182 | 531 | 77
Muscle aches (General disorders) | 254 | 234 | 245 | 733 | 79
Shivering (General disorders) | 92 | 93 | 90 | 275 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.